CLINICAL TRIAL: NCT06533982
Title: Effect of Different Exercise Modalities on Cardiovascular and Cognitive Response in Postmenopausal Women With and Without Vasomotor Symptoms
Brief Title: Effect of Different Exercise Modalities on Cardiovascular and Cognitive Response in Postmenopausal Women
Acronym: WOMEN-EX-MOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Poitiers (Other)
Responsible Party: Principal Investigator, Laurent Bosquet, Director, University of Poitiers
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: WOMEN-EX-MOD
Record Dates: First submitted 2024-07-19; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Menopause; Blood Pressure; Cognitive Decline
Keywords: Physical exercise; High intensity interval exercise; Handgrip
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity interval exercise session (Experimental): Performed on an ergometer, the intensity of the session is adapted to the participant's physical capacity, initially assessed by the VO2max test at baseline.
  The session begins with a 5-minute warm-up at 50% of maximum aerobic power (MAP). The exercise then consists of 2 sets of 12 repetitions of 15 seconds each at 100% of MAP and 15 seconds of passive recovery. 2-minute of passive recovery is recommended between the two sets. The session ends with 5-minute of recovery at 50% of MAP.
  Interventions: Other: High intensity interval exercise session
- Isometric neuromuscular exercise session (Experimental): Performed with a handgrip (K-Force grip, KINVENT), the intensity of the session is adapted to the participant's capacity, initially assessed by the isometric maximal voluntary force (MVF) measurement at the beginning of the session.
  The session consists of 4 repetitions of 2 minutes at 30% of the isometric MVF, separated by 1 minute recovery.
  Interventions: Other: Isometric neuromuscular exercise session
- Control session (No Intervention): Participants are seated for 30 minutes.

INTERVENTIONS:
Other: High intensity interval exercise session — Physical activity session supervised and adapted on ergometer
  Arms: High intensity interval exercise session
Other: Isometric neuromuscular exercise session — Physical activity session supervised and adapted with a handgrip
  Arms: Isometric neuromuscular exercise session

SUMMARY:
Menopause is a natural stage in female aging, increasing cardiometabolic risk and making cardio-neuro-vascular disease (CNVD) the leading cause of mortality in women over 60. Declining ovarian hormones are linked to changes in body composition, increased blood pressure, and mild cognitive impairment. Menopause also often involves significant symptoms like menopausal vasomotor symptoms (VMS), affecting 60-80% of women for 5-10 years. Women with VMS exhibit a worse cardiovascular profile and greater cognitive decline.

Physical exercise is a promising non-pharmacological option to reduce CNVD risk and limit cognitive impairment in postmenopausal women, who have a 10-year window post-menopause during which physical activity benefits vascular and possibly neurovascular health. Studies link physical activity to lower cognitive decline and improved quality of life. However, optimal exercise modalities for managing CNVD risk in postmenopausal women remain undetermined.

DETAILED DESCRIPTION:
Menopause is a natural stage in the female aging process, resulting in increased cardiometabolic risk, making cardio-neuro-vascular disease (CNVD) the leading cause of female mortality worldwide after the age of 60. Indeed, falling ovarian hormone concentrations are associated with altered body composition, increased blood pressure, as well as mild cognitive impairment.

For some women, menopause is also accompanied by symptoms that have a significant impact on their quality of life. Among these, menopausal vasomotor symptoms (VMS - hot flushes, night sweats...) are the most frequent, affecting 60% to 80% of women for an average of 5 to 10 years. Several studies have highlighted an altered cardiovascular profile (dyslipidemia, insulin resistance, pre-hypertension/hypertension...) and a more marked decline in cognitive performance in women with VMS.

In order to reduce the risk of CNVD and limit cognitive impairment, physical exercise appears to be a particularly interesting non-pharmacological management option for postmenopausal women. Indeed, the latter seem to present a 10-year post-menopausal time window, during which physical activity has a positive vascular and probably neurovascular effect, although the latter remains to be demonstrated. Numerous studies have also shown that physical activity is associated with a lower rate of cognitive decline, and improved quality of life.

However, to date, there is little evidence to determine which exercise modalities are most effective in managing the risk of CNVD in postmenopausal women.

The aims of this study:

* To examine the effect of exercise on markers of cardio-neuro-vascular health and cognition in postmenopausal women.
* Second, to compare the differences in the cardio-neuro-vascular and cognitive response to exercise, dependent on the type of exercise, the physical fitness and the presence of menopausal symptoms.
* Third, to examine the effect of menopausal symptoms, and physical fitness on cardio-neuro-vascular health markers and cognitive health markers.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women (absence of menstruation for 12 consecutive months) for less than 10 years
* Women with or without vasomotor symptoms
* Women covered by the French Social Security system

Exclusion Criteria:

* Surgical menopause (oophorectomy)
* Premature ovarian failure
* Chronic renal failure
* Respiratory pathology (unstable asthma, respiratory insufficiency or pulmonary hypertension)
* Cardiovascular disease (coronary, valvular, hypertrophic, hypertensive, infiltrative, constrictive or rhythmic)
* Medically treated hypertension
* Severe obesity (BMI > 40 kg/m²)
* Hearing or vision problems that prevent reading or distinguishing colors
* Recent (< 1 year) central neurological or psychiatric disorders
* Moderate to severe cognitive impairment (MoCA < 18).
* Judicial protection or guardianship

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure (ambulatory blood pressure measurement) | After sessions (24 hours)
  Post-exercise hypotension, using the Mobil-O-Graph (mmHg).
Systolic and diastolic blood pressure (resting) | Before and after sessions (15 minutes)
  Automated oscillometric tensiometer (mmHg).

SECONDARY OUTCOMES:
Concentration of cerebral oxygenation | Before, during, and after sessions (1 hour)
  Near-infrared spectroscopy is used to measure concentrations of oxygenated and desoxygenated hemoglobin (µmol/L).
Working memory | Before and after sessions (10 minutes)
  2-back task (scored from 0 to 28, higher scores indicate better working memory).
Episodic memory | Before and after sessions (15 minutes)
  Memory scale III (MEM-III), a story recall task taken from the test battery in the Wechsler-Memory Scale-Revised (scored from 0 to 25, higher scores indicate better episodic memory).
Executive function | Before and after sessions (15 minutes)
  Stroop task, used to assess inhibitory control (scored as a ratio, negative score indicates worse inhibitory control vs. positive score indicates better inhibitory control).
Perception of exertion | After sessions (1 minute)
  Modified Borg scale (scored 0 to 10, higher score indicates lower exercise tolerance).
Endothelial function (brachial artery dilation capacity) | Baseline (30 minutes)
  At rest, the flow-mediated dilatation technique is used with high-resolution Doppler ultrasound (CX-50 Philipps).
Baroreflex sensitivity | Baseline (1 hour)
  At rest, baroreflex sensitivity is measured using the Finapres.
Aortic systolic and diastolic blood pressure | Baseline (15 minutes)
  At rest, using the SphygmoCor device, which measures central blood pressure (mmHg).
Arterial stiffness (pulse wave velocity) | Baseline (15 minutes)
  At rest, using the SphygmoCor device, which calculates carotid-femoral pulse wave velocity (m/s).
Physical fitness | Baseline (30 minutes)
  Maximal cardiopulmonary effort test (VO2max).
Blood lipid concentrations | Baseline (5 minutes)
  Total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides (g/L).
Blood hormone concentrations | Baseline (5 minutes)
  Progesterone, 17-beta-estradiol, and follicle-stimulating hormone (ng/L).
Body weight | Baseline (1 minute)
  Total body weight, fat mass, fat-free mass and visceral-fat mass in kilograms using the Tanita impedance scale.
Body composition | Baseline (1 minute)
  Percentage of body fat and fat-free mass using the Tanita impedance scale.
Height | Baseline (1 minute)
  Height in meters measured with a height gauge.
Body mass index | Baseline (1 minute)
  Calculated from total body weight and height (kg/m²).
Cognitive assessment | Baseline (15 minutes)
  Montreal Cognitive Assessment (MoCA) test (scored from 0 to 30, with higher scores indicating better cognitive function).
Menopausal rating scale | Baseline (15 minutes)
  Composed of 11 items rating the severity of menopausal symptoms from 0 (no symptoms) to 4 (very severe).
Hot flash related daily interference scale | Baseline (15 minutes)
  Composed of 10 items scored from 0 (no impact) to 10 (completely interferes), evaluating the impact of vasomotor symptoms on daily life.
Hospital Anxiety and Depression Scale | Baseline (15 minutes)
  It provides two scores ranging from 0 to 21 that quantify anxiety and depression. Higher scores indicate more severe symptoms.
Global physical activity questionnaire | Baseline (15 minutes)
  Physical activity and sedentary time assessed using the Global Physical Activity Questionnaire. Higher scores indicate better physical activity levels (categorized into high, moderate, and low physical activity levels).
Daily tobacco and alcohol use | Baseline
  Use daily or not use.
Age | Baseline
  Age, age at menarche and menopause (in years).
Educational level | Baseline
  Secondary education, high school graduate, bachelor's degree, master's or doctoral degree.
Number of children | Baseline
  Self-reported.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bosquet, Pr, Principal Investigator — University of Poitiers - Faculty of Sport Science - MOVE Laboratory (UR20296)
Locations (1):
- Faculty of Sport Science - MOVE Laboratory (UR20296), Poitiers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armas Rojas N, Dobell E, Lacey B, Varona-Perez P, Burrett JA, Lorenzo-Vazquez E, Calderon Martinez M, Sherliker P, Bess Constanten S, Morales Rigau JM, Hernandez Lopez OJ, Martinez Morales MA, Alonso Aloma I, Achiong Estupinan F, Diaz Gonzalez M, Rosquete Munoz N, Cendra Asencio M, Peto R, Emberson J, Duenas Herrera A, Lewington S. Burden of hypertension and associated risks for cardiovascular mortality in Cuba: a prospective cohort study. Lancet Public Health. 2019 Feb;4(2):e107-e115. doi: 10.1016/S2468-2667(18)30210-X. Epub 2019 Jan 23. PMID 30683584
- [Background] Greendale GA, Sternfeld B, Huang M, Han W, Karvonen-Gutierrez C, Ruppert K, Cauley JA, Finkelstein JS, Jiang SF, Karlamangla AS. Changes in body composition and weight during the menopause transition. JCI Insight. 2019 Mar 7;4(5):e124865. doi: 10.1172/jci.insight.124865. eCollection 2019 Mar 7. PMID 30843880
- [Background] Boyle CP, Raji CA, Erickson KI, Lopez OL, Becker JT, Gach HM, Kuller LH, Longstreth W Jr, Carmichael OT, Riedel BC, Thompson PM. Estrogen, brain structure, and cognition in postmenopausal women. Hum Brain Mapp. 2021 Jan;42(1):24-35. doi: 10.1002/hbm.25200. Epub 2020 Sep 10. PMID 32910516
- [Background] Avis NE, Crawford SL, Greendale G, Bromberger JT, Everson-Rose SA, Gold EB, Hess R, Joffe H, Kravitz HM, Tepper PG, Thurston RC; Study of Women's Health Across the Nation. Duration of menopausal vasomotor symptoms over the menopause transition. JAMA Intern Med. 2015 Apr;175(4):531-9. doi: 10.1001/jamainternmed.2014.8063. PMID 25686030
- [Background] Zhu D, Chung HF, Dobson AJ, Pandeya N, Anderson DJ, Kuh D, Hardy R, Brunner EJ, Avis NE, Gold EB, El Khoudary SR, Crawford SL, Mishra GD. Vasomotor menopausal symptoms and risk of cardiovascular disease: a pooled analysis of six prospective studies. Am J Obstet Gynecol. 2020 Dec;223(6):898.e1-898.e16. doi: 10.1016/j.ajog.2020.06.039. Epub 2020 Jun 23. PMID 32585222
- [Background] Gliemann L, Hellsten Y. The exercise timing hypothesis: can exercise training compensate for the reduction in blood vessel function after menopause if timed right? J Physiol. 2019 Oct;597(19):4915-4925. doi: 10.1113/JP277056. Epub 2019 Jun 30. PMID 31077368
- [Background] Anderson D, Seib C, Rasmussen L. Can physical activity prevent physical and cognitive decline in postmenopausal women? A systematic review of the literature. Maturitas. 2014 Sep;79(1):14-33. doi: 10.1016/j.maturitas.2014.06.010. Epub 2014 Jun 20. PMID 25008420
- [Background] Hybholt M. Psychological and social health outcomes of physical activity around menopause: A scoping review of research. Maturitas. 2022 Oct;164:88-97. doi: 10.1016/j.maturitas.2022.07.014. Epub 2022 Aug 3. PMID 35964395
- [Derived] Bourvellec ML, Delpech N, Sosner P, Fritel X, Bosquet L, Enea C. Effect of Exercise Modalities on Post-Exercise Hypotension in Normotensive Postmenopausal Women: A Randomized Controlled Trial on Vasomotor Symptoms Influence. Eur J Sport Sci. 2025 Dec;25(12):e70091. doi: 10.1002/ejsc.70091. PMID 41273313